CLINICAL TRIAL: NCT04934995
Title: Comparison of Arm and Ankle Blood Pressure During Cesarean Delivery: A Blood Pressure Cuffs Pilot Study
Brief Title: Arm and Ankle Blood Pressure Cuffs During C-Section
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ling-Qun Hu, Principal Investigator, Ohio State University
Other Study IDs: 2020H0502
Record Dates: First submitted 2021-03-29; First posted 2021-06-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Supine Hypotensive Syndrome; Cesarean Section Complications; Anesthesia Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: Adult women undergoing cesarean delivery at The Ohio State University Wexner Medical Center under spinal anesthesia, ASA physical status I-III with a BMI during pregnancy ≥ 35 kg/m2 and singleton pregnancy.
  Interventions: Other: Blood Pressure Cuff

INTERVENTIONS:
Other: Blood Pressure Cuff — After obtaining consent and confirming eligibility, Blood Pressure cuffs will be used as specified below:
  Cuff size: large BP cuffs will be the default size for both arm and ankle measurements, but can be changed as clinically indicated based on circumferences of limbs Cuff location: BP cuffs will be placed on the contralateral arm to the main peripheral IV following standard procedures. Left ankle cuff will be placed underneath intermittent pneumatic compression cuffs Ankle blood pressure monitor screen will be covered. Thus, anesthesia providers will not be able to make any clinical decisions based on ankle blood pressures but arm blood pressure (standard) instead.

SUMMARY:
This is a single center prospective self-control study to validate the effectiveness of left uterine displacement after subarachnoid block (SAB) with simultaneous measurements of blood pressure (BP) on the arm and left ankle during surgery in patients undergoing cesarean delivery (CD) at The Ohio State University Wexner Medical Center

DETAILED DESCRIPTION:
In the last three decades, numerous interventions have been studied and implemented into our daily practice, such as pre-loading versus co-loading, phenylephrine versus ephedrine, and phenylephrine infusion versus intermittent boluses. In addition, the effectiveness of left uterine displacement (LUD) to improve blood flow and pressure remains unclear. Also, there are issues to be addressed on this regard, including:

1. Poor placental perfusion from inadequate LUD due to the potential impact of supine hypotensive syndrome (SHS) secondary to aortocaval compression especially after SAB;
2. Shivering during cesarean delivery (CD) resulting in inaccurate BP measurements, the incidence of shivering during CD is reported to be 21.9%. It is unclear the impact of shivering during CD on blood pressure (BP) measurements;
3. Patient discomfort during BP measurements, calf > arm > ankle

The Investigators are conducting a single center prospective self-control study aiming to validate the effectiveness of LUD after SAB with simultaneous measurements of BP on the arm and left ankle during surgery in patients undergoing cesarean delivery (CD). In addition, the Investigators will determine whether ankle BP correlates more accurately than arm SBP with the incidence of nausea/vomiting and category II or III fetal heart tracing and bradycardia after SAB and LUD under no shivering conditions and the impact of body mass index and antepartum estimation of newborn weight on SHS after the SAB.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Women undergoing cesarean delivery at The Ohio State University Wexner Medical Center under spinal anesthesia
3. American Society of Anesthesiologists Physical Status I-III
4. Body mass index during pregnancy ≥ 35 kg/m2
5. Able to consent in English language
6. Singleton pregnancy

Exclusion Criteria:

1. Women undergoing elective cesarean delivery at The Ohio State University Wexner Medical Center under anesthesia other than spinal anesthesia (i.e. general and/or epidural anesthesia)
2. Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women will be included in this study
Study Population: patients undergoing cesarean delivery (CD) at The Ohio State University Wexner Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Difference of SBP measured between arm and ankle during elective CD before SAB | Immediately before subarachnoid anesthesia block (after standard of care left uterine displacement maneuver is performed).
  Arm Systolic Blood Pressure values will be compared with the ankle SBP values before subarachnoid anesthesia. Baseline SBP will be measured pre-spinal anesthesia in supine position (after standard of care left uterine displacement maneuver is performed).
Difference of SBP measured between arm and ankle during elective CD after SAB (before incision) | Immediately after subarachnoid anesthesia block is completed
  Arm Systolic Blood Pressure values will be compared with the ankle SBP values after subarachnoid anesthesia. Postspinal SBP will be measured in supine position, after LUD is performed

SECONDARY OUTCOMES:
Incidence of intraoperative nausea in our patient population | Up to 3 hours from OR admission. Immediately before anesthesia (subarachnoid block) and until operating room discharge
  the incidence of intraoperative nausea will be assessed during anesthesia and surgery
Incidence of intraoperative vomiting in our patient population | Up to 3 hours from OR admission. Immediately before anesthesia (subarachnoid block) and until operating room discharge
  the incidence of intraoperative vomiting will be assessed during anesthesia and surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Qun Hu, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Klohr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta Anaesthesiol Scand. 2010 Sep;54(8):909-21. doi: 10.1111/j.1399-6576.2010.02239.x. Epub 2010 Apr 23. PMID 20455872
- [Background] Hartmann B, Junger A, Klasen J, Benson M, Jost A, Banzhaf A, Hempelmann G. The incidence and risk factors for hypotension after spinal anesthesia induction: an analysis with automated data collection. Anesth Analg. 2002 Jun;94(6):1521-9, table of contents. doi: 10.1097/00000539-200206000-00027. PMID 12032019
- [Background] Bijker JB, van Klei WA, Kappen TH, van Wolfswinkel L, Moons KG, Kalkman CJ. Incidence of intraoperative hypotension as a function of the chosen definition: literature definitions applied to a retrospective cohort using automated data collection. Anesthesiology. 2007 Aug;107(2):213-20. doi: 10.1097/01.anes.0000270724.40897.8e. PMID 17667564
- [Background] Chungsamarnyart Y, Wacharasint P, Carvalho B. Hemodynamic profiles with and without left uterine displacement: A randomized study in term pregnancies receiving subarachnoid blockade for cesarean delivery. J Clin Anesth. 2020 Sep;64:109796. doi: 10.1016/j.jclinane.2020.109796. Epub 2020 Apr 16. PMID 32305794

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT04934995/Prot_SAP_000.pdf